CLINICAL TRIAL: NCT01084928
Title: A Culturally Tailored Lifestyle Intervention to Prevent Diabetes in South Asians
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Diabetes Association (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Venkat Narayan, Hubert Professor of Global Health and Epidemiology, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00035893; 1R34DK081723-01A1 (NIH)
Record Dates: First submitted 2010-03-01; First posted 2010-03-11 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes; Obesity
Keywords: diabetes; obesity; pre-diabetes; South Asian
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Glucose Intolerance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Arm (Diet and Exercise) (Experimental): The lifestyle intervention will include a 16-week intervention period, followed by an 8 week, less intensive maintenance period.
  Interventions: Behavioral: Lifestyle Intervention Classes

INTERVENTIONS:
Behavioral: Lifestyle Intervention Classes — The intervention will be based on the Diabetes Prevention Program but tailored to the needs of the community based on feedback gathered in focus groups. Classes will be group-based and will use a variety of teaching techniques and group-based work to teach participants about behavior change, diet, and physical activity. Participant will be required to attend one group exercise class per week based on traditional Indian dances and other culturally appropriate activities. In order to reach their weekly exercise goal of 150 minutes or more per week, participants will also be able to attend an additional group exercise class, an organized group walk, do a culturally-tailored work out video created by the study staff, and/or exercise on their own.
  Other Names: South Asian Health and Prevention Education (SHAPE)

SUMMARY:
The South Asian Community, people with origins in India, Pakistan, Bangladesh, Maldives, Nepal, Sri Lanka, or Bhutan, are more likely to get diabetes, get diabetes at younger ages, and do worse health-wise once they have diabetes than the general population. This study will test the feasibility and community acceptability of a culturally appropriate lifestyle intervention for the prevention of diabetes in the South Asian community. The outcomes of this project could be used to plan larger interventions to prevent diabetes in South Asians, a rapidly growing segment of the US population.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as being of South Asian origin
* Live in or near Atlanta, Georgia
* BMI greater than 22 kg/m2 calculated from standardized weight and height measurements (a BMI of greater than 22 kg/m2 is indicative of overweight in the South Asian population)
* A confirmed age greater than or equal to 25 determined by checking a valid photo identification (driver's license, passport, etc.)
* No prior diabetes diagnosis (physician diagnosis or on diabetes medication)
* A high risk of developing diabetes (pre-diabetes) as defined by a casual capillary glucose greater than or equal to 120 (measured during screening)
* Fasting glucose of 100-125 mg/dL (impaired fasting glucose tolerance) and/or 2-hour post-load glucose of 140-199 mg/dL (impaired glucose tolerance), measured at baseline visit
* No history of heart disease, serious illness, or conditions that may impede or prohibit participation and are not currently pregnant

Exclusion Criteria:

* Capillary glucose less than 120
* Fasting glucose less than 100 mg/dL or greater than 125 mg/dL OR 2 hour post-load glucose less than 140 mg/dL or greater than 199 mg/dL
* Age less than 25 years
* BMI less than 22 kg/m2
* Pregnancy
* History of heart disease or diabetes (other than gestational diabetes)
* Current functional difficulties
* Severe lung disease or cancer
* Failure to pass cardiovascular stress test

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
body weight | 24 weeks (16 week intervention, 8 week maintenance)

SECONDARY OUTCOMES:
percent body fat | 24 weeks (16 week intervention, 8 week maintenance)
body mass index | 24 weeks (16 week intervention, 8 week maintenance)
waist-to-hip ratio | 24 weeks (16 week intervention, 8 week maintenance)
fasting glucose | 24 weeks (16 week intervention, 8 week maintenance)
blood pressure | 24 weeks (16 week intervention, 8 week maintenance)
plasma lipids | 24 weeks (16 week intervention, 8 week maintenance)
self-reported physical activity | 24 weeks (16 week intervention, 8 week maintenance)
Percent of Total Calories from Fat | 24 weeks (16 week intervention, 8 week maintenance)

CONTACTS AND LOCATIONS:
Overall Officials: Venkat Narayan, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States